CLINICAL TRIAL: NCT00350311
Title: Multicomponent Risk Factor Intervention for People With a Severe Mental Illness: a Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95/05
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Psychotic Disorder; Obesity; Behavior, Addictive
MeSH Terms: conditions — Psychotic Disorders; Obesity; Behavior, Addictive | interventions — Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: nicotine transdermal patch/lozenge

SUMMARY:
This study is a feasibility study of a multi-component intervention to enhance healthy living among young people with psychotic disorders, specifically targeting smoking and weight.

DETAILED DESCRIPTION:
We propose a feasibility study of a multi-component intervention to enhance healthy living among young people (18 to 40 years) with psychotic disorders, specifically targeting smoking and weight. Smoking is very common amongst people with psychotic disorders (around 70% of males, and over 50% of females) and this adds to the overall cardiovascular risk for this group. Obesity is also a common problem for people with psychosis, with an estimated 40-60% being obese or overweight. Obesity in this population may contribute to adverse medical and psychological consequences. For many obese people, targeted pharmacotherapy in addition to diet and increased physical activity can assist in both weight reduction and the maintenance of gains. Similarly, smoking cessation is enhanced by use of adjunctive medications such as nicotine replacement; such strategies continue to produce abstinence rates for up to 10 years.

The proposed study will assess the feasibility of a multi-component behavioural intervention focussing on smoking cessation/diet/physical activity.

The primary outcome measures from the feasibility study are smoking cessation and reduction in body mass index (BMI). Secondary outcomes will include tolerability and safety, as well as the impact the package has on other cardiovascular risk factors including serum lipids, blood sugar levels and depression in young people with psychosis. We will also establish whether smoking cessation and reduction in obesity is correlated with gains in terms of body image, quality and enjoyment of life and reduction in depression. Based on published data, behavioural interventions for smoking cessation and diet and physical activity lead smoking cessation in 20% of people at 12 months and to modest weight loss (around 5%).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 yrs
* DSM-IV diagnosis of non-organic psychotic illness
* Obesity (BMI > 30 or 27 if co-morbidities such as diabetes, hypertension or dyslipidaemia are present
* Current smoker ( > 15 cigarettes per day) if also smoking cannabis regularly, they will still be able to participate

Exclusion Criteria:

* Medical contraindication to exercise or use of the nicotine patch
* Intellectual disability that would significantly impair ability to participate in the program
* Inability to give informed consent (acutely psychotic potential participants will be reassessed one month post screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation
Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Baker, Assoc Prof, Principal Investigator — Centre for Mental Health Studies, Uni of Newcastle
Locations (4):
- Australia (4):
  - Centre for Mental Health Studies, Univeristy Of Newcastle, Newcastle, New South Wales
  - School of Public Health and Community Medicine, University of New South Wales, Sydney, New South Wales
  - Department of Psychiatry, Monash University, The Alfred Hospital, Melbourne, Victoria
  - Mental Health Research Institute, University of Melbourne, Royal Melbourne Hospital, Melbourne, Victoria